CLINICAL TRIAL: NCT06831123
Title: Pathways 2 Success: A Study of School-Based Prevention Programs Supporting Positive Adolescent Development
Brief Title: Pathways 2 Success
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00024346
Record Dates: First submitted 2025-02-07; First posted 2025-02-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Conduct Disorder; Oppositional Defiant Disorder
MeSH Terms: conditions — Conduct Disorder; Oppositional Defiant Disorder | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three different intervention conditions.
Who Masked: Outcomes Assessor
Masking Description: Assessment technicians will not be aware of participants assigned study conditions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Learning to breathe (L2B) (Experimental): randomized to the Learning to Breathe (L2B) mindfulness intervention
  Interventions: Behavioral: L2B
- L2B+App (Experimental): randomized to the Learning to Breathe plus App condition
  Interventions: Behavioral: L2B + App
- Skills for Success (Experimental): randomized to Skills for Success
  Interventions: Behavioral: skills for success

INTERVENTIONS:
Behavioral: L2B — a 6-session, group-based intervention that helps youth develop mindfulness skills
  Arms: The Learning to breathe (L2B)
Behavioral: L2B + App — the Learning to Breathe plus App condition, the 6-session L2B intervention augmented by a mobile application designed to support the use of mindfulness skills in daily life
  Arms: L2B+App
Behavioral: skills for success — a 6-session life skills intervention designed to support decision making and healthy relationships
  Arms: Skills for Success

SUMMARY:
This study involves a 3-arm randomized controlled trial designed to investigate the feasibility and acceptability of three preventive interventions designed to reduce risk for escalations in adolescent conduct problems. High school students identified to be at risk for conduct problems will be randomly assigned to one of three intervention options, including a mindfulness-based program, a mindfulness-based program augmented by a new mobile app, and a life skills program. Assessments related to intervention outcomes will be completed by adolescents, parents/guardians, and teachers at baseline, 2 weeks post-intervention, and at a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. A 9th or 10th grade student in a partner school district
2. Referral due to elevated social/emotional risk indicated on a standardized screening tool or a referral from school support staff due to concerns about school-based conduct problems
3. Adolescents and their parents must be fluent in English

Exclusion Criteria:

1. Currently receiving special education services (i.e., an IEP) due to a behavioral or emotional disturbance
2. Existing diagnoses of autism spectrum disorder, pervasive developmental disorders, developmental/intellectual disability, or serious psychiatric disorders requiring specialized mental health treatment (e.g., psychosis, bipolar, substance use disorder, etc.)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Add Health Self-Report of Delinquency | Baseline; up to 15 weeks; through study completion, approximately 6 months
  A rating scale used to evaluate the number of times in the past month adolescents have committed 17 different antisocial acts.
  A rating scale used to evaluate the number of times in the past month adolescents have committed 17 different antisocial acts. Scores range from 0 to 17, with higher scores reflecting greater engagement in delinquent behaviors.
Behavioral Rating Inventory of Executive Functioning - Second Edition Screening Form | Baseline; up to 15 weeks; through study completion, approximately 6 months
  A 12-item rating scale that evaluates executive functioning A 12-item rating scale that evaluates executive functioning. Scores are reported as T-scores, with higher scores reflecting greater levels of executive functioning difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Piehler, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States